CLINICAL TRIAL: NCT02636283
Title: Use of Entresto (Sacubitril/Valsartan) for the Treatment of Peripheral Arterial Disease
Brief Title: Use of Entresto Sacubitril/Valsartan for the Treatment of Peripheral Arterial Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment
Sponsor: University of Minnesota (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15SDG25360025
Record Dates: First submitted 2015-10-29; First posted 2015-12-21 (Estimated); Results first posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Entresto (Active Comparator): oral route
  Interventions: Drug: Entresto
- Placebo group (Placebo Comparator): Oral placebo
  Interventions: Drug: Placebo group

INTERVENTIONS:
Drug: Entresto — Oral pills
  Arms: Entresto
Drug: Placebo group — The placebo pills
  Arms: Placebo group

SUMMARY:
This study proposes the use of Entresto (sacubitril/valsartan) to test the effects on pain free walking duration on patients with peripheral arterial disease, a condition caused by decreased blood flow to the muscles in the legs.

DETAILED DESCRIPTION:
Current approaches for the treatment of peripheral arterial disease (PAD) lack the success observed in the treatment of other forms of vascular diseases. A potential reason for this may be that available treatments do not target the pathological mechanisms implicated in the development of PAD. These mechanisms include obstruction of aortic-iliac arteries and its branches due to the formation of atherosclerotic plaques and mitochondrial and microvascular dysfunction. Although blood flow improves following surgical revascularization, pain free and maximal walking duration does not improve to the same degree. This suggests that in addition to blood flow obstruction, mitochondrial and microvascular dysfunction are significant factors implicated in the development of PAD.

Therefore, any treatment designed for patients with PAD should be aimed at improving mitochondrial and microvascular function. In this regard, natriuretic peptides (NP) have been shown to increase mitochondrial and microvascular density and these two findings have been associated with increases in oxygen consumption and perfusion of skeletal muscles.

The Investigator proposes that an increase in endogenous natriuretic peptides by inhibiting the enzyme that degrades it in blood will increase mitochondrial and microvascular function and this will be associated with an increase in maximal and pain free walking duration. To test this hypothesis the investigators have designed a double blind randomized controlled clinical trial providing sacubitril/valsartan for 12 weeks trial period.The improvements in mitochondrial and microvascular function will be measured using magnetic resonance (MR) spectroscopy and functional MR imaging and an exercise stress test will be used to assess maximal and pain free walking duration. This trial will provide patients with PAD with a non-surgical, cause-specific treatment option.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with symptoms of intermittent claudication, such as exercise-induced pain, cramps, fatigue, or other equivalent discomfort, involving large muscle groups of the leg(s) (calf, thigh, buttocks), relieved by rest.
2. Ankle-brachial index ≤ 0.90 acquired according to the American Heart Association guidelines.
3. Highest ankle pressure reduced by at least 25 mm Hg after exercise compared to resting pressure (or loss of previously present Doppler signal for both the posterior tibial and anterior tibial arteries immediately after exercise if arteries were incompressible).
4. Patients on medical treatment for PAD without significant improvement in intermittent claudication within the last 6 months.

Exclusion Criteria:

1. Age < 18 and > 80 years.
2. Patients with physician diagnosed chronic kidney disease or heart failure stage II or IV or unstable angina.
3. Echocardiographic evidence of cardiomyopathies and pulmonary hypertension.
4. Patients that have received cancer treatment within the last year (except skin cancer).
5. Severe limitations in mobility due to osteomuscular disorders present at time of interview.
6. Dementia or other mental disorders that prevent patients from following a research protocol present at time of interview
7. Patients engaged in an exercise rehabilitation program within the past 6 months.
8. Patients schedule to undergo an arterial revascularization procedure during the study or have undergone one within the past 6 months.
9. Inconsistent maximal walking distance on the treadmill test.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-12-31 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Otto A Sanchez, M.D., Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Entresto | Placebo Group
Started | 3 | 3
Completed | 1 | 0
Not Completed | 2 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Trial Terminated Prematurely | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Entresto | Placebo Group | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (4.16) | 62.7 (3.06) | 61.7 (3.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 00 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Treadmill Walk Until Pain Initiated in Minutes
Description: Time in minutes on a standardized treadmill test to initiation of pain and time until pain requires patient to stop walking
Time Frame: 12 weeks
Population: Study terminated prematurely; outcome measure data was not collected.
Arm/Group | Entresto | Placebo Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Mitochondrial and Microvascular Function Arterial Elasticity
Description: Post-contraction measures of mitochondrial and microvascular function using MR spectroscopy and functional MRI
Time Frame: 12 weeks
Population: Study terminated prematurely; outcome measure data was not collected.
Arm/Group | Entresto | Placebo Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Insulin Sensitivity
Description: Using Homeostasis Model Assessment (HOMA) index
Time Frame: 12 weeks
Population: Study terminated prematurely; outcome measure data was not collected.
Arm/Group | Entresto | Placebo Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Arterial Elasticity
Description: Pulse wave pressure analysis
Time Frame: 12 weeks
Population: Study terminated prematurely; outcome measure data was not collected.
Arm/Group | Entresto | Placebo Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Quality of Life Questionnaires
Description: Questionnaires describing independent living and quality of life
Time Frame: 12 weeks
Population: Study terminated prematurely; outcome measure data was not collected.
Arm/Group | Entresto | Placebo Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Entresto | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entresto (N=3) | Placebo Group (N=3)
Chest Discomfort (General disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) — Pain during study procedure due to pre-existing condition

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT02636283/Prot_SAP_000.pdf